CLINICAL TRIAL: NCT03543319
Title: Norwegian Microemboli in Acute Stroke Study (NOR-MASS)
Brief Title: Norwegian Microemboli in Acute Stroke Study
Acronym: NOR-MASS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Other Study IDs: REK 2018/589
Record Dates: First submitted 2018-05-11; First posted 2018-06-01 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2018-06

CONDITIONS: Ischemic Stroke; Embolic Stroke; Microemboli
MeSH Terms: conditions — Ischemic Stroke; Embolic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
BACKGROUND: The cause of ischemic stroke remains undetermined in 30-40% of the cases, but circulating blood clots (thromboemboli) are a postulated common denominator in approx. 75% of patients. Transcranial Doppler monitoring (TCDM) is a non-invasive method of detecting circulating microemboli (CME) in the human cerebral circulation. The method is not used systematically in unselected groups of patients with repeated long-term registrations. New ultrasound equipment is ambulatory, less unpleasant for the patient and allows extended monitoring sessions. This may vastly simplify the implementation of TCDM as a clinically useful diagnostic tool.

AIMS: Determine the usefulness of TCDM in acute stroke diagnostics by assessing prevalence and frequency of CME in unselected patients with ischemic stroke, the influence of antithrombotic drugs on CME and the relationship between MES and recurrent stroke or transient ischemic attack (TIA).

HYPOTHESES: Prevalence and frequency of CME are higher during the first 24 hours than at later follow-up. Stroke etiology can be assessed by the presence or absence of CME. Presence of CME is associated with increased risk of recurrent TIA of stroke within 3 months and 1 year. Cessation of CME after the start of antithrombotic treatment is associated with reduced risk of recurrent TIA or stroke.

DETAILED DESCRIPTION:
* Standardized questionnaire
* Clinical work-up in accordance with hospital standard operating procedures, i.e. radiological and cardiological procedures, neurovascular ultrasound, clinical scoring, etc.
* 1st Transcranial Doppler monitoring (TCDM) at admission if within 24 hours after stroke onset (day 1). TCDM is repeated at 18-36 hours and at day 3. Microembolic signals are automatically registered by the software and subsequently verified manually.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to hospital < 24 hours after onset of ischemic stroke

Exclusion Criteria:

* Temporal bone window inadequate for transcranial Doppler examination
* Participation in ongoing sonothrombolysis study (NOR-SASS 2)
* Reduced ability to cooperate
* No informed consent can be obtained

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke or TIA admitted to Haukeland University Hospital. All stroke sub-types, severities and vascular distributions are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-06-12 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of circulating microemboli | Up to 24 hours after symptom onset

SECONDARY OUTCOMES:
Prevalence of circulating microemboli as a function of time and antithrombotic drugs | 3 days after symptom onset
Prevalence of MRI DWI lesions | 18-36 hours after symptom onset
Recurrence of ischemic stroke/TIA | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Derived] Aarli SJ, Thomassen L, Logallo N, Kvistad CE, Naess H, Fromm A. Prolonged and repeated microemboli detection in acute ischemic stroke - The Norwegian Microemboli in Acute Stroke Study (NOR-MASS). J Stroke Cerebrovasc Dis. 2024 Sep;33(9):107849. doi: 10.1016/j.jstrokecerebrovasdis.2024.107849. Epub 2024 Jul 5. PMID 38972617